CLINICAL TRIAL: NCT00650546
Title: Role of Exenatide in Treatment of NASH-a Pilot Study
Brief Title: Role of Exenatide in NASH-a Pilot Study
Acronym: NAFLD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DK61737; U01DK061737 (NIH)
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Non-alcoholic steatohepatitis; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A pre treatment NAS score (Experimental): liver biopsy score pre treatment with exenatide 5 micrograms SQ (sub-cutaneous) twice a day titrated to 10 mcg SQ twice a day as tolerated
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 5 mcg twice a day titrated to 10 mcg twice a day
  Other Names: Byetta

SUMMARY:
We hypothesize that exenatide (Byetta), a GLP-1 agonist administered subcutaneously for 24-28 weeks improves liver histology in diabetic patients with biopsy-proven NASH.

DETAILED DESCRIPTION:
Eight adult patients with known type 2 DM(Diabetic) and biopsy-proven NAFLD were treated with 5-10 mcg subcutaneous exenatide for 28 weeks. Liver histology was assessed using the NAFLD Activity Score (NAS) prior to therapy and after 28 weeks of therapy. We used the following criteria to define our primary outcome: (i) no worsening of fibrosis score, (ii) improved score by at least one point in hepatocyte ballooning, (iii) either (a) improvement in NAS by 2 or more points spread across at least two of the three NAS components, or (b) post-treatment NAS equal or greater than 3.

ELIGIBILITY:
Inclusion Criteria:

* Well documented NASH based on clinical and histological criteria. Liver biopsy must have been obtained within 12-months prior to initiation of the study.
* Subjects must have known diabetes (either diet controlled or only on Metformin or sulfonylureas such as glyburide or glipizide).
* Subjects must be 18 year or older.

Exclusion Criteria:

* Co-existing etiologies for chronic liver disease (hepatitis B or C, autoimmune or hemochromatosis, etc.).
* Clinical or histological evidence of cirrhosis.
* Alanine aminotransferase or aspartate aminotransferase > 300 IU/L.
* Uncontrolled diabetes (hemoglobin A1C greater than or equal to 9%).
* Insulin or TZD dependant DM.
* Known human immunodeficiency virus infection.
* Current or history of significant alcohol consumption within past 5 years. Significant alcohol consumption is defined as >20 grm/day in females and >30 grms/day in males or if alcohol consumption cannot satisfactorily be quantified.
* Serum creatinine of greater than or equal to 2 mg/dl.
* Active, serious medical disease (cardiac, renal, pulmonary, dermatologic, psychiatric illness) with likely life expectancy less 5 years.
* Current or previous malignancy with expected life expectancy less than 5-years (other than basal cell cancer of the skin).
* Use of drugs historically associated with NASH.
* Histological evidence of malignancy, 4+ iron deposition, or any other type of liver disease.
* Active substance abuse, such as alcohol,inhaled or injection drugs with the previous one year.
* Known intolerance or allergy to exenatide (Byetta).
* History of neuroglycopenia.
* Women of childbearing potential must have had a negative pregnancy test prior to starting the study and should be willing to avoid pregnancy during the study period.
* Women must not be nursing.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naga Chalasani, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Indiana University, Indianapolis, Indiana
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Fort Sam Houston, San Antonio, Texas

REFERENCES:
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Younossi ZM, Gramlich T, Matteoni CA, Boparai N, McCullough AJ. Nonalcoholic fatty liver disease in patients with type 2 diabetes. Clin Gastroenterol Hepatol. 2004 Mar;2(3):262-5. doi: 10.1016/s1542-3565(04)00014-x. PMID 15017611
- [Background] Kolterman OG, Buse JB, Fineman MS, Gaines E, Heintz S, Bicsak TA, Taylor K, Kim D, Aisporna M, Wang Y, Baron AD. Synthetic exendin-4 (exenatide) significantly reduces postprandial and fasting plasma glucose in subjects with type 2 diabetes. J Clin Endocrinol Metab. 2003 Jul;88(7):3082-9. doi: 10.1210/jc.2002-021545. PMID 12843147
- [Background] Promrat K, Lutchman G, Uwaifo GI, Freedman RJ, Soza A, Heller T, Doo E, Ghany M, Premkumar A, Park Y, Liang TJ, Yanovski JA, Kleiner DE, Hoofnagle JH. A pilot study of pioglitazone treatment for nonalcoholic steatohepatitis. Hepatology. 2004 Jan;39(1):188-96. doi: 10.1002/hep.20012. PMID 14752837
- [Background] Shadid S, Jensen MD. Effect of pioglitazone on biochemical indices of non-alcoholic fatty liver disease in upper body obesity. Clin Gastroenterol Hepatol. 2003 Sep;1(5):384-7. doi: 10.1053/s1542-3565(03)00198-8. PMID 15017657
- [Background] Neuschwander-Tetri BA, Brunt EM, Wehmeier KR, Oliver D, Bacon BR. Improved nonalcoholic steatohepatitis after 48 weeks of treatment with the PPAR-gamma ligand rosiglitazone. Hepatology. 2003 Oct;38(4):1008-17. doi: 10.1053/jhep.2003.50420. PMID 14512888
- [Background] Eng J, Andrews PC, Kleinman WA, Singh L, Raufman JP. Purification and structure of exendin-3, a new pancreatic secretagogue isolated from Heloderma horridum venom. J Biol Chem. 1990 Nov 25;265(33):20259-62. PMID 1700785
- [Background] Eng J, Kleinman WA, Singh L, Singh G, Raufman JP. Isolation and characterization of exendin-4, an exendin-3 analogue, from Heloderma suspectum venom. Further evidence for an exendin receptor on dispersed acini from guinea pig pancreas. J Biol Chem. 1992 Apr 15;267(11):7402-5. PMID 1313797
- [Background] Chen YE, Drucker DJ. Tissue-specific expression of unique mRNAs that encode proglucagon-derived peptides or exendin 4 in the lizard. J Biol Chem. 1997 Feb 14;272(7):4108-15. doi: 10.1074/jbc.272.7.4108. PMID 9020121
- [Background] Greig NH, Holloway HW, De Ore KA, Jani D, Wang Y, Zhou J, Garant MJ, Egan JM. Once daily injection of exendin-4 to diabetic mice achieves long-term beneficial effects on blood glucose concentrations. Diabetologia. 1999 Jan;42(1):45-50. doi: 10.1007/s001250051111. PMID 10027577
- [Result] Kenny PR, Brady DE, Torres DM, Ragozzino L, Chalasani N, Harrison SA. Exenatide in the treatment of diabetic patients with non-alcoholic steatohepatitis: a case series. Am J Gastroenterol. 2010 Dec;105(12):2707-9. doi: 10.1038/ajg.2010.363. No abstract available. PMID 21131943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 recruitment sites: Department of Gastroenterology, San Antonio Uniformed Services Health Consortium, San Antonio, Texas, USA. Indiana University School of Medicine, Indianapolis, IN, USA
Pre-assignment Details: This was a single arm, open label study. Only study group received exenatide treatment. Eight adult patients with known type 2 DM and biopsy-proven NAFLD were treated with 5-10mcg subcutaneous exenatide for 28 week.All eight patients were started on exenatide 5 mcg injections twice a day and the dose was increased to 10 mcg injections twice a day
Groups:
- Exenatide Group: Exenatide 5 micrograms SQ twice a day titrated to 10 mcg SQ twice a day as tolerated
  Exenatide : 5 mcg twice a day titrated to 10 mcg twice a day
Period: Overall Study
Arm/Group | Exenatide Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: eight adult patients with known type 2 DM and biopsy -proven NAFLD were treated with 5-10 subcutaneous exenatide for 28 weeks
Groups:
- Open-labeled Prospective Case Series: Exenatide 5 micrograms SQ twice a day titrated to 10 mcg SQ twice a day as tolerated
  Exenatide: 5 mcg twice a day titrated to 10 mcg twice a day
Arm/Group | Open-labeled Prospective Case Series
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54 [36 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Number of participants who had NAFLD Activity Score (NAS) pre/post 24-28 wks. after treatment [Number; unit: participants] — The NAFLD Activity Score (NAS) is an underweight sum of steatosis (score 0-3), inflammation (score 0-3), ballooning scores (0-2). The NAS can range from 0-8 with the higher score indicating more aggressive disease.
  participants | 8
NAS score [Median (Full Range); unit: units on a scale] — steatosis, inflammation, ballooning. Each catagory has a 1 to 3 value given and the total of all 3 catagories equals the NAS overall score. 1] The NAFLD Activity Score (NAS) is an underweight sum of steatosis (score 0-3), inflammation (score 0-3), ballooning scores (0-2). The NAS can range from 0-8 with the higher score indicating more aggressive disease
  units on a scale | 4 [3 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Improvement in Liver Histology After Treatment With Exenatide
Description: Number of patients with liver histology improved with exenatide. The improvement of liver histology was defined as (1) no worsening of the fibrosis score, (11) improved score by at least one point in hepatocyte ballooning, and (111) either (a) improvement in NAS (NAFLD Activity Score) by two points spread across as least two of the three NAS components, or by (B)post-treatment NAS<3.
Time Frame: between baseline and 24-28 weeks after initiating treatment
Measure: Number; unit: participants
Groups:
- Treatment With Exenatide: eight adult patients with known type 2 DM and biopsy proven NAFLD
Arm/Group | Treatment With Exenatide
Number analyzed (Participants) | 8
participants | 8

2. Primary Outcome: Change in NAS
Description: The NAFLD Activity Score (NAS) is an underweight sum of steatosis (score 0-3), inflammation (score 0-3), ballooning scores (0-2). The NAS can range from 0-8 with the higher score indicating more aggressive disease.
Time Frame: Between baseline and 28 weeks of treatment with exenatide, sub q, 5-10 mcq.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Individuals Who Recieved Treatment With Exenatide: change of NAS score in eight adult patients with known type 2 DM and biopsy proven NAFLD after treatment with exenatide
Arm/Group | Individuals Who Recieved Treatment With Exenatide
Number analyzed (Participants) | 8
units on a scale | -1.5 (1.66)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Exenatide Group
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Group (N=8)
abdominal pain along with nausea (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
As a case series our findings are limited by a control group and a small number of subjects enrolled. These limitations are tempered by the single expert hepatologist and the stringent definitions for histological improvement, ((primary end point)..

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No